CLINICAL TRIAL: NCT05153668
Title: AERO: Adjuvant EveRolimus Outcomes in Laryngotracheal Stenosis
Brief Title: Everolimus Trial in Laryngotracheal Stenosis
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00284589
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Subglottic Tracheal Stenosis
Keywords: Tracheal Stenosis; Everolimus; Immunosuppression
MeSH Terms: conditions — Idiopathic subglottic tracheal stenosis; Tracheal Stenosis | interventions — Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adjuvant Everolimus After Surgical Dilation (Experimental): Individuals will take low dose everolimus for 6 weeks after dilation.
  Interventions: Drug: Everolimus Oral Tablet

INTERVENTIONS:
Drug: Everolimus Oral Tablet — Everolimus 1.5mg by mouth daily will be given for 42 days after dilation surgery.
  Other Names: Zortress

SUMMARY:
Subglottic stenosis (obstructing scar in the larynx and trachea) occurs in patients spontaneously (idiopathic), with autoimmune disease, and after long-term breathing tube placement and can result in communication disability and high mortality rates due to the obstructed airway. The proposed Adjuvant EveRolimus Outcomes (AERO) trial is proof-of-concept study using the immunosuppressant drug, everolimus, to reduce the number of surgeries for patients with idiopathic Subglottic Stenosis (iSGS). Success with the AERO trial will allow for everolimus to be used in subsequent larger trials of participants with laryngotracheal stenosis and could lead to everolimus being the first FDA approved medical treatment for iSGS.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of laryngotracheal stenosis
* Patient age 18 - 80 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Serum total bilirubin and Serum Glutamic Pyruvic Transaminase (SGPT)/(ALT) < 2.0 times the upper limit of normal;
* Serum creatinine < 2.0 mg/dL;
* The patient must be able to comprehend and have signed the informed consent.
* The patient must have documentation of their date of laryngotracheal stenosis diagnosis and prior medical/surgical history.
* Participants must have also had a prior suspension microlaryngoscopy with endoscopic excision of scar and balloon dilation procedure prior to study entry

Exclusion Criteria:

* Use of corticosteroids (glucocorticoids) within 7 days of everolimus administration (except physiologic dose equivalent)
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within 7 days of registration
* Participation in any clinical trial within 21 days of bone marrow collection involving an investigational drug or device
* History of malignancy within five years of registration, except adequately treated basal or squamous cell skin cancer
* History of an autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus) requiring active systemic treatment. Hypothyroidism without evidence of Grave's disease or Hashimoto's thyroiditis is permitted.
* Human T-cell Lymphotropic Virus type 1 (HTLV-1) or type 2 (HTLV-2)
* New York Heart Association (NYHA) class II-IV heart failure within the past 6 months
* History of organ transplant with use of immunosuppression
* Current use of immunosuppression
* Contraindication or documented intolerance to everolimus
* Women of childbearing potential who are not on highly effective contraception or abstinent for at least 30 days. Highly effective contraception includes at least two forms of concurrent contraception (Condoms, oral contraceptives, intrauterine devices, contraceptive implants).
* Women who are pregnant or breastfeeding, or wishing to become pregnant are excluded from this study
* Current use of cytochrome P450 3A inducers (such as some anticonvulsants, rifampin, isoniazid, St. John's wort).
* Current use of cytochrome P450 3A inhibitors (such as azole antifungals, nondihydropyridine calcium channel blockers, some macrolide antibiotics, grapefruit) can result in significant interactions
* Baseline proteinuria as defined by urine dipstick analysis
* History of angioedema
* Baseline/continued use of drugs known to be associated with angioedema including angiotensin converting enzyme inhibitors
* Significant pulmonary disease independent of laryngotracheal stenosis as defined by and forced expiratory volume at one second (FEV1)/forced vital capacity (FVC) < 10% of the expected value for the patient's age.
* Evidence of a COVID-19 infection including anosmia, upper respiratory symptoms or positive test result within the 30 days prior of trial participation.
* Patients who are not fully vaccinated for COVID 19 for at least 4 weeks prior to study entry
* Immunosuppressive therapy within previous 21 days or expected need for immunosuppressive therapy for the duration of the study
* Known immunodeficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Expiratory flow in patients with Laryngotracheal Stenosis | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 1 year, 2 years
  Change in Peak Expiratory flow (L/min) in patients with Laryngotracheal Stenosis will be assessed.

SECONDARY OUTCOMES:
Dilation interval (time between surgery) | Up to 2 years
  Dilation interval (time between surgery) in months will be assessed.
Change in Voice-related Quality of Life Score | Baseline, 1 month, 2 months, 3 months, 6 months, 1 year, 2 years
  Number scale of 0-100
Change in Clinical Chronic Obstructive Pulmonary Disease (COPD) Questionnaire Quality of Life Score | Baseline, 1 month, 2 months, 3 months, 6 months, 1 year, 2 years
  Number scale of 0-6
Change in Eating Assessment Tool (EAT-10) Swallow Quality of Life Score | Baseline, 1 month, 2 months, 3 months, 6 months, 1 year, 2 years
  Number scale of 0-40
Change in 12-Item Short Form (SF-12) Survey Global Quality of Life Score | Baseline, 1 month, 2 months, 3 months, 6 months, 1 year, 2 years
  Number scale of 0-100
Change in lumen surface area | Baseline and 6 months
  CT Neck will be used to assess change in lumen surface area in millimeters squared (mm^2).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hillel, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] So RJ, Collins SL, Collins S, Mafla L, Chan-Li Y, Lina I, Gelbard A, Motz KM, Hillel AT. Oral Everolimus Following Dilation in Idiopathic Subglottic Stenosis: A Phase 1 Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2024 Nov 1;150(11):1029-1033. doi: 10.1001/jamaoto.2024.2886. PMID 39325463